CLINICAL TRIAL: NCT04356300
Title: Exosome of Mesenchymal Stem Cells for Multiple Organ Dysfuntion Syndrome After Surgical Repaire of Acute Type A Aortic Dissection: a Pilot Study
Brief Title: Exosome of Mesenchymal Stem Cells for Multiple Organ Dysfuntion Syndrome After Surgical Repaire of Acute Type A Aortic Dissection
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Liang-Wan Chen MD, Department Director, Fujian Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020005
Record Dates: First submitted 2020-04-19; First posted 2020-04-22 (Actual); Last update posted 2020-05-06 (Actual); Status verified 2020-05

CONDITIONS: Multiple Organ Failure
MeSH Terms: conditions — Multiple Organ Failure

STUDY DESIGN:
Intervention Model Description: Part 1: totally 30 patient will be enrolled, and 15 patients will be given Exosomes of MSCs immediately after ascending aortic replacement combined with open placement of triple-branched stent graft for ATAAD.
  Part 2: totally 30 patient will be enrolled, and 15 patients will be given Exosomes of MSC after onset of multiple organ dysfuntion syndrome after ascending aortic replacement combined with open placement of triple-branched stent graft for ATAAD.
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The exosome of MSC arm (Experimental): Exosome of MSC at a dose of 150mg will be given intravenously to Patients in the exosome of MSC arm once a day for 14 times.
  Interventions: Biological: Exosome of MSC
- The control arm (No Intervention): Patients in the control arm will not be given exosome of MSC.

INTERVENTIONS:
Biological: Exosome of MSC — Exosome of MSC at a dose of 150mg will be given intravenously to patients once a day for 14 times.
  Arms: The exosome of MSC arm

SUMMARY:
Multiple organ dysfunction syndrome (MODS) after surgical repaired for acute type A aortic dissection (ATAAD) is a life-threatening condition. In this study, patients who undergoing surgical repaired of ATAAD immediately or presenting sever MODS after surgical repaired of acute type A aortic dissection will be treated with umbilical cord-derived mesenchymal stem cell.

DETAILED DESCRIPTION:
Multiple organ dysfunction syndrome (MODS) are common debilitating complications after surgical repaired for ATAAD. MODS is one of the chief causes of post-operative death for acute type A aortic dissection (ATAAD) patients, and it was reported that MODS accounted for more than half of the death after surgery for ATAAD. Despite recent advance in surgical technique, mortality rate remains high in such critical care conditions. In animal models, studies have demonstrated the beneficial effects of MSCs with respect to ischemia-reperfusion injury of heart, lungs, kidney, brains and livers. Several pilot studies have provided evidence that MSC may be effective in treating critically ill patients with traumatic brain injury, acute renal failure, or acute respiratory distress syndrome. There is increasing evidence that MSCs function in a paracrine manner. Exosomes have been reported to activate signaling pathways by binding to receptors. Compared with mesenchymal stem cells, exosomes are more stable and storable and no risk of aneuploidy. The possibility of immune rejection after allogeneic administration of exosomes is lower and can provide alternative treatment for a variety of diseases.

The trial contains two parts:

Part one (prevention scheme):to explore the safety and efficacy of exosome of MSC, the investigators will recruit patients who are diagnosed with ATAAD, and 15 participants will be administrated intravenously with exosome of MSC immediately after ascending aortic replacement combined with open placement of triple branched stent graft while other 15 not. Then the investigators will monitor participants' MODS related biochemical indexes, sequential organ failure assessment (SOFA) scores, comparing to those don't be treated with exosome of MSC.

Phase two (treatment scheme): for patients presenting severe MODS (SOFA score≥10) after ascending aortic replacement combined with open placement of triple-branched stent graft, the investigators will randomly use exosome of MSC to 15 of participants while other 15 not. Then the investigators will monitor participants' MODS related biochemical indexes, SOFA scores, comparing to those don't be treated with MSC. The dosage of the exosome of MSC was determined on the basis of the previous clinical studies, which is 180mg once a time and administrated intravenously.

ELIGIBILITY:
Inclusion Criteria:

* Part 1:

  * Patients who are diagnosed with ATAAD and received emergency surgery with ascending aortic replacement combined with open placement of triple-branched stent graft
  * elder than 60 years old
  * Preoperative PaO2/FiO2 ≥ 400mmHg, platelets ≥ 150*109/L, bilirubin≥ 20μmol/L, no hypotension (without vasoactive drugs), Glasgow Coma Score Scale = 15, creatine ≥110μmol/L

Part 2:

* Patients who are diagnosed with ATAAD and received emergency surgery with ascending aortic replacement combined with open placement of triple-branched stent graft
* Patients who have failure of at least 2 organs
* Patients who meet the criteria as below:

sequential organ failure assessment score (SOFA) ≥ 10

Exclusion Criteria:

* • uncontrollable underlying disease life expectancy of less than 4 days history of long-term corticosteroid use during the past 6 months.

  * The pre-operative computer tomography angiography(CTA) demonstrate the visceral arteries are involved
  * pre-existing severe disease of any major organs

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2021-09-01 (Estimated); Study Completion 2030-09-01 (Estimated)

PRIMARY OUTCOMES:
survival after intervention | Up to 6 month
  comparing survival ratio in hospital(6 months post-intervention) between groups.
sequential organ failure assessment score | Up to 6 months
  Compare the change of sequential organ failure assessment score between groups. Scores ranged from 0 to 24. The higher the score, the worse the prognosis.
interleukin-6 | Early 3 days
  Compare the change of concentration of interleukin( IL)-6 between groups.
The number of allergic reactions | Up to 6 months
  Allergic reactions are mostly manifested as skin flushing, rash and itching. Severe allergic reactions such as chills, high fever and anaphylactic shock are rare.
The number of people who get cancer | Up to 2 years
  The number of people diagnosed with cancer after treatment

SECONDARY OUTCOMES:
the effects on kidney function | Up to 6 months
  the therapeutic effects in the improvement of kidney function, as indicated by Scr level.
the effects on liver function | Up to 6 months
  the therapeutic effects in the improvement of liver function, as indicated by bilirubin levels.
the effects on lung function | Up to 6 months
  the therapeutic effects in the improvement of lung function, as indicated by oxygenation index.
the effects on coagulation function | Up to 6 months
  the therapeutic effects in the improvement of coagulation function, as indicated by blood platelet count.
the effects on central nervous system | Up to 6 months
  The Glasgow coma scale has a maximum score of 15 and a minimum score of 3, indicating consciousness. 12-14 was classified as mild consciousness disorder; 9-11 was classified as moderate disturbance of consciousness; A score below 8 is coma; The lower the score, the greater the disturbance of consciousness.

CONTACTS AND LOCATIONS:
Overall Officials: Liang-wan Chen, M.D, Principal Investigator — Union Hospital

IPD SHARING:
Plan to Share IPD: No